CLINICAL TRIAL: NCT01389206
Title: Pulmonary Arterial Hypertension Quality Enhancement Research Initiative Extension Program
Acronym: PAH QuERI Ext
Status: Completed | Type: Observational
Sponsor: Actelion (Industry)
Collaborators: Canadian Heart Research Centre (Other)
Responsible Party: Sponsor
Other Study IDs: AC-052-428
Record Dates: First submitted 2011-07-06; First posted 2011-07-08 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Observation; Bosentan; Iloprost; Epoprostenol

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Standard of care: Observational study to improve the management of PAH patients through an evidence-based approach aimed at achieving optimal WHO functional class (FC) treated with Tracleer, Ventavis, Veletri, Opsumit and/or Uptravi.
  Interventions: Drug: observational study with patients treated with Tracleer, Ventavis, Veletri, Opsumit and/or Uptravi

INTERVENTIONS:
Drug: observational study with patients treated with Tracleer, Ventavis, Veletri, Opsumit and/or Uptravi — observational study with patients treated with Tracleer, Ventavis, Veletri, Opsumit and/or Uptravi

SUMMARY:
Knowledge Translation Program for the guidelines and evidence-based management of PAH patients

DETAILED DESCRIPTION:
To improve the management of PAH patients through an evidence-based approach aimed at achieving optimal WHO functional class (defined as: 1) improvement of FC III or IV to FC II; 2) improvement of FC II to FC I; or 3) maintaining FC II or I)

ELIGIBILITY:
Inclusion Criteria:

1. Male and female adults (≥ 18 years of age)
2. Documented diagnosis of PAH (all of the following): i. RHC demonstrating mPAP > 25 mm Hg and PCWP

   ≤ 15 and PVR > 3 ii. FEV 1 > 50% predicted normal iii. V/Q and/or CT scan excluding the thromboembolic etiology
3. Diagnosis of PAH < 3 years
4. Need for PAH specific treatment
5. Desire to participate and signs an informed consent

Exclusion Criteria:

Any of the criteria below:

1. Poor mental function, drug or substance (e.g.,alcohol) abuse, or unstable psychiatric illness, which, in the opinion of the investigator, may interfere with optimal participation in the study
2. Prior participation in this program
3. Patients with pulmonary hypertension classified as group 2 - 5 Updated Clinical Classification of Pulmonary Hypertension (5th World Symposium on PH Modified Classification of PH)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 800 PAH patients from approximately 80 physician practices will be included in the program.
Sampling Method: Non-Probability Sample
Enrollment: 797 (Actual)
Dates: Start 2011-06-01; Primary Completion 2018-04-10 (Actual); Study Completion 2018-04-10 (Actual)

PRIMARY OUTCOMES:
Patients achieving guideline-recommended treatment | 3 years
  Proportion of patients achieving guideline-recommended treatment

SECONDARY OUTCOMES:
Patients achieving optimal functional class | 3 years
  Proportion of patients achieving optimal functional class using an evidence-based treatment algorithm

CONTACTS AND LOCATIONS:
Overall Officials: Vallerie McLaughlin, MD, Study Chair — University of Michigan
Locations (76):
- United States (75):
  - Cardiovascular Associates, PC, Birmingham, Alabama
  - University of South Alabama Medical Center, Mobile, Alabama
  - Pulmonary Associates, Phoenix, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Alliance Medical and Research Center, Fountain Valley, California
  - Scripps Clinic, Scripps Green Hospital, La Jolla, California
  - University of Southern California, Los Angeles, California
  - Paloma Medical Group, San Juan Capistrano, California
  - Harbor-UCLA Medical Center, Torrance, California
  - University of Colorado Denver, Aurora, Colorado
  - South Denver Cardiology Associates PC, Littleton, Colorado
  - Robert E. Benkert, M.D.P.C., Wheat Ridge, Colorado
  - Lung Health & Sleep Enhancement Center, LLC, Newark, Delaware
  - Bay Area Cardiology Research, P.A., Brandon, Florida
  - Bay Area Chest Physicians, Clearwater, Florida
  - Broward Pulmonary and Sleep Specialists, Fort Lauderdale, Florida
  - Pulmonary Diseases, Internal Medicine, Critical Care Medicine, Fort Lauderdale, Florida
  - Mount Sinai Medical Centre - Columbia University - Division of Cardiology, Miami Beach, Florida
  - Central Florida Pulmonary Group, PA, Orlando, Florida
  - Lung Associates of Sarasota, Sarasota, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - University of Illinois at Chicago, Chicago, Illinois
  - Unity Point Health Pulmonary Services, Peoria, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - Kentuckiana Pulmonary Associates, Louisville, Kentucky
  - University of Louisville School of Medicine, Louisville, Kentucky
  - Ochsner Medical Center, New Orleans, Louisiana
  - Maine Medical Center, Portland, Maine
  - University of Maryland Medical Centre, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - University of Michigan Pulmonary Hypertension Program, Ann Arbor, Michigan
  - Wayne State University, Detroit Medical Center, Detroit, Michigan
  - Spectrum Health, Grand Rapids, Michigan
  - William Beaumont Hospital - Troy, Troy, Michigan
  - Nebraska Pulmonary Specialties, LLC, Lincoln, Nebraska
  - Creighton University Medical Centre - Pulmonary, Critical Care and Sleep Medicine Division, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - The Lung Center of Nevada, Las Vegas, Nevada
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Michael Schwarz, MDFACC, Bloomfield, New Jersey
  - Respiratory Health & Critical Care Associates, Hawthorne, New Jersey
  - Pulmonary Hypertension & Lung Transplant Program Newark Beth Israel Medical Center, Newark, New Jersey
  - North Shore - LIJ Health System, New Hyde Park, New York
  - Beth Israel Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University Phyisicans Clinic/Pulmonary, Winston-Salem, North Carolina
  - The Christ Hospital Heart & Vascular Center, Cincinnati, Ohio
  - University of Cincinnati Pulmonary Critical Care & Sleep Medicine, Cincinnati, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Dayton Respiratory Center, Dayton, Ohio
  - University of Toledo Health Sciences Campus, Toledo, Ohio
  - Heart Center Cardiology, Bend, Oregon
  - Central Bucks Specialists - The Pavilion at Doylestown Hospital, Doylestown, Pennsylvania
  - Institute for Respiratory and Sleep Medicine, Langhorne, Pennsylvania
  - Pulmonary Hypertension Program, Cardiology, Children's Hospial of Philadelphia, Philadelphia, Pennsylvania
  - Pulmonary Vascular Disease Program, Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Respiratory Specialists, Wyomissing, Pennsylvania
  - Wellspan Lung, Sleep and Critical Care, York, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Sioux Falls Cardiovascular PC, Sioux Falls, South Dakota
  - Statcare Pulmonary Consultants, Knoxville, Tennessee
  - El Paso Respiratory and Sleep Consultants, El Paso, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Baylor College of Medicine, Houston, Texas
  - UT Health - University of Texas Houston, Houston, Texas
  - Providence Health Center, Waco, Texas
  - IHVI, Advanced Lung Disease and Transplant Clinic, Falls Church, Virginia
  - Sentara Medical Group, Norfolk, Virginia
  - Cardiac Study Center, Puyallup, Washington
- PAH Clinic CPR at Auxilio Mutuo, San Juan, Puerto Rico